CLINICAL TRIAL: NCT01700595
Title: Preexpanded Perforator Flaps in Pediatric Patients
Brief Title: Preexpanded Perforator Flaps in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Emre Hocaoglu, Specialist, M.D., Istanbul University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: hocaoglupediatricperforator1; emrehocaoglu (Registry Identifier: clinical trials)
Record Dates: First submitted 2012-10-01; First posted 2012-10-04 (Estimated); Last update posted 2012-10-04 (Estimated); Status verified 2012-10

CONDITIONS: Contractures; Scars
MeSH Terms: conditions — Contracture; Cicatrix

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- new technical intervention (Experimental): ''new technical intervention'' represents the surgical procedure which is applied for the patients assigned to this group because of their certain characteristics. Namely, pediatric patients with broad axillary, anterior chest wall, mammary and neck scars are treated with this surgical approach.
  Interventions: Procedure: new technical intervention

INTERVENTIONS:
Procedure: new technical intervention — Contractures and broad scars of the subjects are treated by this surgical intervention which is a reconstructive surgery that is performed by the transfer of preexpanded perforator flaps to the recipient sites of skin deficiency.
  Other Names: reconstructive surgery by transfer of preexpanded perforator flaps

SUMMARY:
Contractures and broad scars of the axilla, anterior chest wall and neck have detrimental effects on functional, physical and psychological development of children. Perforator flaps have already been shown to be reliable options for the reconstruction of contractures but there have been no reports demonstrating the value of preexpanded perforator flaps of dorsolateral trunk region in treatment of extensive contractures and scars of pediatric patients. The purpose of this study is to demonstrate these techniques by a case series formed of pediatric patients with broad scars and contractures of anterior chest wall, axilla, neck and breasts. Seven pediatric patients (mean age, 11,6 years) who were treated by preexpanded perforator flaps are presented. By this means, clinical experience on intercostal artery perforator (ICAP) flap, thoracodorsal artery perforator (TDAP) flap, circumflex scapular artery perforator (CSAP) flap and lumbar artery perforator flap was shared. Flaps as large as 20,5x10,5 cm in size could be successfully transferred in pediatric patients. Broad scar tissues were resurfaced with broad flaps carrying similar characteristics with the uninjured anterior chest wall and neck skin in six of our patients. In one patient with partial necrosis, full thickness skin graft was used for the residual defect. The mean duration of postoperative (after flap transfer) follow-ups was 17,2 months. The preexpanded TDAP, ICAP and CSAP flaps are revealed to be useful reconstructive options for the treatment of scars and contractures of anterior chest wall, axilla, neck and breast in pediatric patients.

ELIGIBILITY:
Inclusion Criteria:

* pediatric age group
* broad scars and contractures

Exclusion Criteria:

* age over 18 years
* minimal scars and skin defects that could be treated by minor interventions

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 7 (Actual)
Dates: Start 2012-09; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Range of motion of the particular joint | at least three months after flap tarnsfer
  Disruption of the contracture band and releasing the contracture of a particular joint results in achievement of the healthy range of motion of that joint.

SECONDARY OUTCOMES:
Replaced tissue dimensions | at least three months after the operation
  Transferred flap sizes will be documented. It is a way of demonstrating the amount of replaced scar tissue and exhibiting the success of the technique.

OTHER OUTCOMES:
Developement of related anatomic structures | at least a year after flap transfer
  Resurfacing the broad scar tissue and releasing the contracture leads to normal developement of the relevant extremity, chest, neck, breast and posture of the patient, thus, providing the healthy developement of the child.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul University, Istanbul Faculty of Medicine, Istanbul, Turkey (Türkiye)

REFERENCES:
- [Derived] Hocaoglu E, Aydin H. Preexpanded perforator flaps of the dorsolateral trunk in pediatric patients. Plast Reconstr Surg. 2013 May;131(5):1077-1086. doi: 10.1097/PRS.0b013e3182865dd7. PMID 23385985